CLINICAL TRIAL: NCT05565794
Title: A Phase II Study of Pemigatinib After Curative Local Therapy in Locally Advanced Intrahepatic Cholangiocarcinoma (iCCA) Harboring FGFR2 Fusions/Rearrangements.
Brief Title: Pemigatinib After Curative Local Therapy in Advanced iCCA With FGFR2 Fusion/Rearrangements
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEARLDIFER; 2021-006232-50 (EudraCT Number); IKF-t055 (Other: IKF Trial ID)
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma; FGFR2 Gene Mutation; FGFR2 Gene Rearrangement; FGFR2 Gene Translocation
Keywords: intrahepatic cholangiocarcinoma; iCCA; FGFR2 fusion; FGRF2 rearrangement; FGFR2 alteration; FGFR2 mutation
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pemigatinib (Experimental): Intake of 13.5 mg pemigatinib once daily per oral
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Intake of up to 3 tablets of pemigatinib (4,5 mg each) daily per oral for 14 days in a 21-day cycle (maximum of 18 cycles in total)
  Other Names: Pemazyre

SUMMARY:
The aim of this phase II study is to determine whether pemigatinib is clinically efficious after curative local therapy such as surgery/ SBRT or ablation in iCCA patients harboring FGFR2 fusion/rearrangement and to assess the safety profile to support the continuation of the concept in a large, randomized trial for further development.

DETAILED DESCRIPTION:
This is a prospective, exploratory, single-arm, non-randomized, open-label phase II study to investigate whether pemigatinib is clinically efficacious after curative local treatment including surgery/ SBRT or ablation in iCCA patients with FGFR2 fusion/rearrangements.

Patients will receive pemigatinib 13.5 mg oral once daily (21-day cycle; two weeks on, one week off) until disease recurrence, unacceptable toxicity, withdrawal of consent, or investigator decision, but no longer than 12 months (max. 18 cycles).

The primary objective is to assess the efficacy of pemigatinib administered after curative local therapy in treatment-naïve patients with resectable intrahepatic biliary tract cancer (recurrence free survival rate at 12 months, RFS@12).

Secondary objectives are to assess the efficacy by overall survival (OS) and recurrence free survival (RFS); to assess safety of the treatment (AEs, impact on liver function, use of subsequent therapies); to assess quality of life (QoL).

In addition, tissue samples will be analyzed for biomarkers predictive for RFS and OS.

20 patients are to be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for trial participation:

* Signed informed consent form (ICF).
* Patients*, age ≥ 18 years at the time of signing the informed consent form.
* Histologically proven and curatively treatable localized intrahepatic biliary tract cancer (iCCA only) with a previous maximum of 5 cm in diameter, without signs of metastatic disease, and proven FGRF2- fusions/ rearrangements, identified by routine FISH or by NGS testing.

Note: Only CE-IVD marked NGS-tests are applicable which cover FGFR2 fusions and rearrangements

* Patients previously received SBRT or another minimally invasive technique (e.g., laparoscopic liver resection) up to 12 weeks prior to enrolment
* Female patients who are considered as woman of childbearing potential (WOCBP) as well as male patients who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment as well as up to 1 week after the last dose of pemigatinib. Female patients who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile, see section 13.5) as well as azoospermic male patients do not require contraception. Female patients considered as WOCBP must have a negative pregnancy test within the last 7 days prior to the start of study therapy.
* ECOG performance status 0-1.
* Appropriate hematological, hepatic and renal function:

  1. Absolute number of neutrophils ≥ 1.5 x 109/L
  2. Platelets ≥ 100 x 109/L
  3. Hemoglobin ≥ 9 g/dL (5.58 mmol/L)
  4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  5. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN without existing liver metastases, or ≤ 5 x ULN in the presence of liver metastases; AP ≤ 5 x ULN.
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance (measured by 24h urine) ≥ 40 mL/min (i.e., if the serum creatinine level is > 1.5 x ULN, then a 24-h urine test must be performed to check the creatinine clearance to be determined).
* Adequate coagulability, as determined by the International Normalized Ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 5 s above the ULN (unless anti-coagulation therapy has been given). Patients receiving warfarin / Phenoprocoumon must be switched to low molecular weight heparin before starting any study-specific procedures.
* Patients must be able to take oral medications.
* For patients with active hepatitis B virus (HBV):

HBV DNA ≤ 500 IU/mL obtained within 28 days prior to initiation of study treatment, AND Anti-HBV treatment (per local standard of care e.g. entecavir) prior to study entry and willingness to continue treatment for the length of the study.

- For patients with active hepatitis C virus (HCV): Patients positive for HCV antibody are eligible, also if polymerase chain reaction testing is positive for HCV RNA However, anti-viral therapy against HCV is only allowed prior to trial but not during the trial.

* Patients infected with human immunodeficiency virus (HIV) are eligible if they meet all the following criteria:

  1. CD4 count is ≥350 cells/uL, viral load is undetectable, and not taking prohibited cytochrome (CYP)-interacting medications
  2. Probable long-term survival with HIV if cancer were not present
  3. Stable on a highly active antiretroviral therapy (HAART) regimen for ≥4 weeks and willing to adhere to their HAART regimen with minimal overlapping toxicity and drug-drug interactions with the experimental agents in this study
  4. HIV is not multi-drug resistant
  5. Taking medication and/or receiving antiretroviral therapy that does not interact or have overlapping toxicities with the study medication
* Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment, and scheduled visits and examinations including follow up.

Exclusion Criteria:

Patients who meet at least one of the following criteria are not eligible for trial participation:

* Presence of tumors other than biliary tract cancer or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. The Sponsor decides to include patients who have received curative treatment and have been disease-free for at least 3 years.
* Metastatic biliary tract cancer (intrahepatic, hilar, or distal CCA as well as gallbladder carcinoma) disease.
* Pretreatment with any systemic anti-cancer therapy.
* Simultaneous, ongoing systemic immunotherapy, chemotherapy, or hormone therapy not described in the study protocol.
* Simultaneous treatment with a different anti-cancer therapy other than that provided in the study (excluding palliative radiotherapy only for symptom control).
* Previous therapy with an FGFR- inhibitor.
* Stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
* Known allergic / hypersensitive reactions to at least one of the treatment components.
* Other serious illnesses or medical ailments within the last 12 months prior to the start of the study.
* Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to central serous retinopathy, macular/retinal degeneration, diabetic retinopathy, retinal detachment) as confirmed by ophthalmologic examination.
* History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues, such as the skin, kidney, tendons or vessels due to injury, disease, and aging, in the absence of systemic mineral imbalance).
* History of hypovitaminosis D requiring supraphysiologic doses (eg, 50,000 UI/weekly) to replenish the deficiency. NOTE: Participants receiving vitamin D supplements are eligible .
* Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study treatment. NOTE: Moderate CYP3A4 inhibitors are not prohibited (refer to section Fehler! Verweisquelle konnte nicht gefunden werden. Appendix 3 for a list of CYP3A4 inhibitors and inducers).
* Presence of an active, uncontrollable infection.
* Has active infection with SARS-CoV-2 (positive antigen test in routine testing at site).
* Chronic inflammatory bowel disease.
* Active disseminated intravascular coagulation.
* Any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
* On-treatment participation in another interventional clinical study in the period 30 days prior to inclusion and during the study.
* Patient pregnant or breast feeding, or planning to become pregnant
* Patient in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4).
* Subjects that are depending on the Sponsor/CRO or investigational site as well as on the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate at time of progression | through study completion, approx. 3 years
  Objective response rate according to investigator-based RECIST 1.1 assessment, defined as the proportion of allocated subjects with best response of complete or partial response within 12 months after the date of first administration of study treatment. Patients who receive anti-cancer treatment other than the study medication for any reason before reaching a complete or partial response will be identified as nonresponders in the assessment of ORR.

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  Overall survival until end of study
Quality of Life asssed by EORTC-QLQ-C30 with additional appendix BIL21 | from screening until end of study, approx. 3 years
  Measurement of quality of life by questionaires filld in by the patients.
Incidence of treatment-related adverse events | from screening until end of study, approx. 3 years
  Safety and tolerability will by measured by evaluation of incidence, treatment relationship, seriousness, and severity of all AEs, SAEs according to CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Goetze, Prof. Dr., Principal Investigator — Krankenhaus Nordwest, Frankfurt; Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH
Locations (10):
- Germany (10):
  - Universitätsklinikum Augsburg III. Medizinische Klinik, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln AöR Klinik für Gastroenterologie und Hepatologie, Cologne
  - Medizinische Klinik und Poliklinik I Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf
  - Klinikum Esslingen GmbH Klinik für Allgemeine Innere Medizin Onkologie / Hämatologie, Gastroenterologie und Infektiologie, Esslingen am Neckar
  - Klinikum Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Jena Klinik für Innere Medizin II, Jena
  - TUM Universitätsklinikum Klinikum rechts der Isar Technische Universität München Klinik für Poliklinik und für Innere Medizin, München

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.